CLINICAL TRIAL: NCT00299663
Title: Long Term Follow-up of Patients With Group A Streptococcal Infection Originating From the Genital Tract
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Ahinoam Lev-Sagie, MD, Hadassah Medical Organization
Other Study IDs: GAS-HMO-CTIL
Record Dates: First submitted 2006-03-05; First posted 2006-03-07 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Streptococcal Infections
Keywords: group A streptococcal infection; genital tract; CARRIER; patients with GAS isolation; Streptococcus Group A
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Group A streptococcus (GAS) causes a variety of human infections. It is also an uncommon but serious cause of postpartum infections. In contrast to group B streptococcus (GBS) infection, which causes illness and death in newborns disproportionately more often than it does in mothers, perinatal GAS infection primarily affects mothers . Invasive GAS infection is defined by the isolation of GAS from a normally sterile site (e.g., blood) or by the isolation of GAS from a nonsterile site in the presence of the streptococcal toxic shock syndrome or necrotizing fasciitis. A postpartum case of invasive GAS is defined as isolation of GAS during the postpartum period, in association with a clinical postpartum infection (e.g., endometritis) or from either a sterile site or a wound infection.

Because of the burden and severity of invasive GAS infection, the Centers for Disease Control and Prevention (CDC) hosted a meeting in to formulate guidelines for responding to postpartum and postsurgical GAS infections. However, we could not find any recommendations for long-term follow-up of patients who had GAS infection subsequent to delivery or gynaecological procedures, or further recommendations regarding subsequent delivery or gynaecological invasive procedures. It is possible that women who had GAS as a cause of vaginal infection may have a tendency to be carriers of this organism, but this has never been proven. We believe it is of importance to determine if women who have had one infection may be long-term carriers which may pose a risk during future pregnancies.

The objective of the present study is to evaluate the incidence of long term gynaecological carrier state of patients who had GAS invasive infection following delivery, and to provide guidelines for follow-up and treatment of such patients.

The proposed study may answer the question whether this endogenous GAS origin represents chronic GAS carrier state, similar to the known GBS carrier state. As some of these patients had severe infections (sometimes life threatening) a protocol for long-term follow up and management is necessary in case an invasive procedure is done (IUD insertion, endometrial biopsy, curettage or delivery) in order to prevent recurrent infection. The information collected in the study will enable us to afford recommendations for follow up and prophylaxis in the future.

.

DETAILED DESCRIPTION:
Research plan The study population will include patients diagnosed with GAS invasive infection following delivery or gynaecological procedures (such as endometrial biopsy, D&C or IUD insertion) at Hadassah university hospitals, and patients in whom an isolation of GAS from the vagina without infection was reported. The study will consist of two parts, prospective and retrospective.

1. Retrospective study

   1. The records of all patients diagnosed with GAS infection/isolation in the past 3 years (2003-2005) will be reviewed. The estimated occurrence of GAS isolation from the genital tract in Hadassah hospital is 15 cases every year (Moses personal communication).
   2. Patients' files will be reviewed for demographic and clinical variables associated with the development of GAS infection (age, parity, obstetric history), its clinical course and subsequent progress to septic shock, and the site of GAS isolation (blood, vaginal discharge, wound etc).
   3. Additional information will be obtained from the patients in order to evaluate the incidence of gynaecological infections and risk factors for such infections. These include events of pelvic inflammatory disease, contraceptive methods, subsequent deliveries or D&C (a questionnaire is attached).
   4. Vaginal cultures and pharyngeal swabs will be taken from all women with previous gynecological GAS infection/isolation participating in the study, in order to evaluate whether carriage of GAS in the vagina occurs.
2. emm typing Since we have the original isolates from women with invasive disease (those presenting with bacteremia) we will be able to compare the specific type isolate obtained in consequent cultures with the original isolate. Isolates will be compared by several known bacterial attributes such as emm type, T type, and the presence of genes for the different exotoxins. emm typing PCR of streptococcal isolates will be performed as previously described [11], according to the recommendations of the Division of Bacterial and Mycotic Diseases, Streptococcus pyogenes emm sequence database (http://www.cdc.gov/ncidod/biotech/strep/doc.htm).
3. Prospective study- In addition to the above patients, women presenting from the beginning of the study for two years, with an isolation of GAS from the vagina (even without overt disease), will be followed in order to evaluate the significance of such isolates. These isolates will be collected for comparison with surveillance cultures which will be taken in the future. Vaginal cultures and pharyngeal swabs will be taken every 2 months during the year.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with GAS infection/isolation in the past 3 years (2003-2005)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population that participate in the study are women who were udentified with positive culture of group A streptoccoci in the genital tracts, starting from 2003 and on.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2006-02; Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLON MOSES, Study Director — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] 1. Chuang I, Van Beneden C, Beall B, Schuchat A. Population-based surveillance for postpartum invasive group a streptococcus infections, 1995-2000. Clin Infect Dis. 2002:15;35:665-70. 2. Centers for Disease Control and Prevention. Active bacterial core surveillance (ABCs) report: group A Streptococcus, 2000. 3. The Working Group on Severe Streptococcal Infections. Defining the group A streptococcal toxic shock syndrome. Rationale and consensus definition. JAMA 1993; 269:390 1. 4. Stevens DL, Tanner MH, Winship J, et al. Severe group A streptococcal infections associated with a toxic shock like syndrome and scarlet fever toxin A. N Engl J Med 1989; 321:1 7. 5. Centers for Disease Control and Prevention. Case definitions for infectious conditions under public health surveillance. MMWR Recomm Rep 1997;46(RR-10):1 55. 6. Prevention of Invasive Group A Streptococcal Infections Workshop Participants .Prevention of invasive group A streptococcal disease among household contacts of case patients and among postpartum and postsurgical patients: recommendations from the Centers for Disease Control and Prevention. Clin Infect Dis. 2003 15;36:243.